CLINICAL TRIAL: NCT04849182
Title: Randomized, 3-arm Controlled Clinical Trial, Designed to Evaluate the Effectiveness of Supplementation With Vertistop® D and Vertistop® L in Preventing Recurrence of High-recurrence BPPV (Benign Paroxysmal Positional Vertigo)
Brief Title: Vertistop® D and Vertistop® L in Preventing Recurrence of High-recurrence BPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Locale di Matera (Other)
Responsible Party: Principal Investigator, Prof. Giacinto Asprella Libonati, Medical Executive, Azienda Sanitaria Locale di Matera
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VERT-2017-001
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Benign Paroxysmal Positional Vertigo (BPPV)
Keywords: BPPV; Vertistop; Vitamin D; Alpha-lipoic acid; Zinc
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vertistop D (Active Comparator): Patients with deficiency (<20 ng/mL, <50 nmol/L) or insufficiency (20-30 ng/mL, 50-75 nmol/L) of Vitamin D
  Interventions: Dietary Supplement: Vertistop D
- Vertistop L (Active Comparator): Patients with normal vitamin D levels (>30 ng/mL, >75 nmol/L)
  Interventions: Dietary Supplement: Vertistop L
- Control group (No Intervention): Patients meeting the inclusion criteria with normal levels of vitamin D (>30 ng/mL, >75 nmol/L)

INTERVENTIONS:
Dietary Supplement: Vertistop D — Food supplement containing alpha-lipoic acid, carnosine, zinc, vitamin D3 and vitamins of group B, 1 tablet/day before meals
  Arms: Vertistop D
Dietary Supplement: Vertistop L — Food supplement containing alpha-lipoic acid, carnosine, zinc and curcumin, 2 tablets/day (morning and evening)
  Arms: Vertistop L

SUMMARY:
Randomized, 3-arm controlled clinical study, to evaluate the effectiveness of supplementation with Vertistop® D (food supplement containing alpha-lipoic acid at modified release, Carnosine and Zinc, Vitamin D and Vitamins B) and Vertistop® L (food supplement containing fast releasing alpha-lipoic acid, Carnosine, Zinc and Curcumin) in preventing recurrence of high-recurrence BPPV (Benign Paroxysmal Positional Vertigo)

DETAILED DESCRIPTION:
Benign paroxysmal positional vertigo (BPPV) is the most common type of vertigo detectable in otoneurological clinical practice. It is characterized by violent, short and relapsing vertiginous crises that arise when the patient assumes certain positions of the head in the space and is accompanied by a usually "typical" paroxysmal positional nystagmus. In most cases we cannot trace the exact causal agent, so we mainly identify two forms: primitive forms and secondary forms. BPPV therapy is essentially physical, and it is based on specific maneuvers which make the otoconial mass come out of the semicircular canal. Recent studies showed the existence of a seasonal trend of BPPV related to fluctuations in Vitamin D levels. Based on these considerations this clinical trial was designed in order to evaluate the possible efficacy of the administration of Vitamin D (Vertistop® D) in preventing recurrence of BPPV.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary BPPV;
* Patients having BPPV of CSP or CSL (geo or apo, single or multi channel);
* Patients with recurrent BPPV, defined as two or more episodes over the last six months, or three or more episodes in the last 12 months;
* Informed consent.

Exclusion Criteria:

* Patients under 18 years of age;
* Secondary BPPV;
* Vitamin D levels greater than 100 ng/mL (>250 nmol/L);
* Pregnant or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Number of BPPV recurrences in patients supplemented with Vertistop D | 0, 6 months
  Change in the number of BPPV recurrences associated with the increase or normalization of Vitamin D serum levels after supplementation with Vertistop D

SECONDARY OUTCOMES:
Number of BPPV recurrences in patients supplemented with Vertistop-L | 0, 6 months
  This parameter is defined as the difference in the number of BPPV recurrences observed in the period between the baseline visit and the final visit (after 6 months)
Mean difference in Dizziness Handicap Inventory (DHI) values | 0, 6 months
  This parameter is defined as the mean difference in the DHI values between the baseline visit and the final visit (after 6 months)
Mean difference in the Visual Numeric Scale (VNS) values | 0, 6 months
  This parameter is defined as the mean difference in the VNS values between the baseline visit and the final visit (after 6 months)
Mean difference in the Visual Analogue Scale (VAS) values | 0, 6 months
  This parameter is defined as the mean difference in the VAS values between the baseline visit and the final visit (after 6 months)

OTHER OUTCOMES:
Incidence of adverse events | 2, 4, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Policoro Hospital "Giovanni Paolo II", Matera, Italy